CLINICAL TRIAL: NCT05093296
Title: Oxytocin and Naltrexone: Investigation of Combined Effects on Stress- and Alcohol Cue-induced Craving in Alcohol Use Disorder - a Randomized Double-blind Placebo-controlled Parallel-group Trial
Brief Title: Oxytocin and Naltrexone: Investigation of Combined Effects on Stress- and Alcohol Cue-induced Craving in Alcohol Use Disorder
Acronym: ON-ICE
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Central Institute of Mental Health, Mannheim (Other)
Collaborators: Heidelberg University - Institute of Medical Biometry (IMBI) (Unknown); Heidelberg University - Coordination Centre for Clinical Trials (KKS) of Heidelberg University (Unknown); German Federal Ministry of Education and Research (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CIMH ON-ICE 21
Record Dates: First submitted 2021-10-13; First posted 2021-10-26 (Actual); Last update posted 2024-03-29 (Actual); Status verified 2024-03

CONDITIONS: Alcohol Use Disorder; Alcoholism; Alcohol Addiction
MeSH Terms: conditions — Alcoholism | interventions — Naltrexone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oxytocin + Naltrexone (Experimental): All patients will receive 50mg Naltrexone daily (NTX, oral tablet) in the course of standard in-patient treatment. In the experimental group, patients will receive a single dose of 24 I.U. oxytocin nasal spray at two study visits during in-patient treatment:
  * Visit 2 - First Application of Oxytocin 40 minutes prior to a combined stress- and alcohol cue-exposure during visit 2
  * Visit 3 - Second Application of Oxytocin 40 minutes prior to an fMRI-based assessment of alcohol cue-reactivity
  Interventions: Drug: Oxytocin nasal spray; Drug: Naltrexone Pill
- Placebo + Naltrexone (Active Comparator): All patients will receive 50mg Naltrexone daily (NTX, oral tablet) in the course of standard in-patient treatment. In the comparator group, patients will receive a placebo nasal spray (same composition as the verum oxytocin spray except for the active ingredient oxytocin) at two study visits during in-patient treatment:
  * Visit 2 - First Application of Placebo 40 minutes prior to a combined stress- and alcohol cue-exposure during visit 2
  * Visit 3 - Second Application of Placebo 40 minutes prior to an fMRI-based assessment of alcohol cue-reactivity
  Interventions: Drug: Naltrexone Pill; Drug: Placebo

INTERVENTIONS:
Drug: Oxytocin nasal spray — 24 I.U. Oxytocin nasal Spray will be administered twice on two separate trial days.
  Arms: Oxytocin + Naltrexone
Drug: Naltrexone Pill — All participants will receive 50mg Naltrexone daily as oral tablet throughout the study
Drug: Placebo — Placebo nasal spray (same composition as the verum oxytocin spray except for the active ingredient oxytocin)
  Arms: Placebo + Naltrexone

SUMMARY:
Alcohol use disorder (AUD) is a chronic relapsing disorder. Alcohol craving, a hallmark symptom of AUD that drives relapse in patients, is only insufficiently treated by existing medication. One promising new compound is Oxytocin (OXY), which showed beneficial effects on alcohol craving in preliminary clinical studies. Additionally, OXY seems to enhance effects of established medication, specifically Naltrexone (NTX), an opioid-antagonist which is approved for AUD treatment via positive synergism on neurotransmitter levels. The proposed two-armed, 1:1 randomized, double-blind, parallel group trial seeks to test the putative synergistic effects of combined intranasal OXY spray (24 IU) + oral NTX (50mg) against Placebo spray + oral NTX (50mg) on alcohol craving (primary outcome) in male and female patients with AUD that suffer from high alcohol craving, within the framework of a validated alcohol cue-and stress-exposure task (i.e. a combined Trier Stress Test and alcohol cue-exposure) that was established for screening new medications in AUD and determine their effects on craving and relapse risk. Treatment effects on additional neurobiological and biochemical markers of craving that show strong associations to individual relapse risk, will serve as secondary outcomes. Collection and analysis of follow-up data (90 days) will be performed to determine whether treatment effects relate to patient outcome.

The clinical trial period for an individual participant consists of a screening visit (visit 1), a baseline visit (visit 2) and two treatment visits (visits 3 and 4)(all within equal or less than ten days) followed by a 90 days (+/- 7 days) follow-up phase with two visits (visits 5 and 6) at day 30 (± 7 days) and day 90 (± 7 days). Visits 1 to 4 will be conducted while participants are undergoing standard in-patient treatment at the Department of Addictive Behavior and Addiction medicine at the Central Institute of Mental Health (CIMH) in Mannheim, Germany, for the medical condition under investigation.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 70 years
* Patients meeting the diagnosis of an alcohol dependence according to the Internation Clasification of Diseases 10th revision (ICD10)
* Patients with at least moderate craving, i.e. either >=15 points on the Alcohol Urge Questionnaire (AUQ, range 8 to 56 points) craving scale or increase in AUQ scores by >= 50% after exposure to visual alcohol cues (i.e. minimum increase of >=4 points after cue exposure)
* Ability of the individual to understand the character and the individual consequences of the clinical trial
* Written informed consent (must be available before enrollment in the study)
* Consent to random assignment
* For women with childbearing potential, use of a highly effective birth control method until 24 hours after Visit 4 and negative pregnancy test

Exclusion Criteria:

* Subjects presenting with any of the following criteria will not be included in the clinical trial: Current psychotic or bipolar disorder or current severe depressive episode with suicidal ideations
* Current treatment with any of the following substances: Any investigational medicinal product, Opioid-containing Analgesics, Anorexics, Anticonvulsants, Opioid-containing Antidiarrheal Agents, Antineoplastics, Antipsychotics (exception: episodic use of melperone, pipamperone and quetiapine are allowed), Antidepressants (exception: allowed, when being taken in stable dose for a minimum of 14 days prior to enrolment and/or doxepin in low doses [max. 75mg daily]), Opioid-containing Cough/cold agents, systemic Steroids
* Positive drug screening (amphetamines/ecstasy, opiates, cocaine, barbiturates)
* Pregnancy, lactation or breastfeeding
* Current severe somatic comorbidities: liver cirrhosis [CHILD B or C] or impaired renal function [glomerular filtration rate (GFR)<15ml/Min] [each determined by physical examination and/or laboratory testing], severe heart insufficiency [determined by assessment of medical history], pre-existing epilepsy [determined by assessment of medical history], long-QT syndrome or cardial arrhythmia [determined by ECG]
* History of hypersensitivity to the investigational medicinal product Oxytocin (Syntocinon®) and/or Naltrexone (trade names: Adepend, Naltrexon-Hcl neuraxpharm, Naltrexonhydrochlorid Accord) or to any drug with similar chemical structure or to any excipient present in the pharmaceutical form of the investigational medicinal product Oxytocin (Syntocinon®) and/or Naltrexone
* Participation in other clinical trials or observation period of competing clinical trials, respectively.
* Acute suicidal tendency or acute endangerment of self and others

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2021-12-02 (Actual); Primary Completion 2023-07-15 (Actual); Study Completion 2023-09-27 (Actual)

PRIMARY OUTCOMES:
Alcohol Urge Questionnaire (AUQ) | 60 minutes after oxytocin/placebo application and directly after the combined stress- and cue-exposure will serve as primary outcome measure at Visit 3
  Subjective Alcohol Craving will be assessed at separate time points before and after Oxytocin Administration using the AUQ

SECONDARY OUTCOMES:
Alcohol Urge Questionnaire (AUQ) | 35 minutes after oxytocin/placebo application at Visit 3
  Subjective Alcohol Craving will be assessed at separate time points before and after Oxytocin Administration using the AUQ
Alcohol Urge Questionnaire (AUQ) | 70 minutes after oxytocin/placebo application at Visit 3
  Subjective Alcohol Craving will be assessed at separate time points before and after Oxytocin Administration using the AUQ
Alcohol Urge Questionnaire (AUQ) | 80 minutes after oxytocin/placebo application at Visit 3
  Subjective Alcohol Craving will be assessed at separate time points before and after Oxytocin Administration using the AUQ
Alcohol Urge Questionnaire (AUQ) | 90 minutes after oxytocin/placebo application at Visit 3
  Subjective Alcohol Craving will be assessed at separate time points before and after Oxytocin Administration using the AUQ
Alcohol Urge Questionnaire (AUQ) | 85 minutes after oxytocin/placebo application, i.e. directly fMRI session at Visit 4
  Subjective Alcohol Craving will be assessed at separate time points before and after Oxytocin Administration using the AUQ
Primary Appraisal secondary Appraisal Scale (PASA) | 35 minutes after oxytocin/placebo application at Visit 3
  Perceived stress will be assessed using the Primary Appraisal secondary Appraisal Scale (PASA) at separate time points before and after Oxytocin Administration using the AUQ at Visit 3 and Visit 4
Primary Appraisal secondary Appraisal Scale (PASA) | 60 minutes after oxytocin/placebo application at Visit 3
  Perceived stress will be assessed using the Primary Appraisal secondary Appraisal Scale (PASA) at separate time points before and after Oxytocin Administration using the AUQ at Visit 3 and Visit 4
Primary Appraisal secondary Appraisal Scale (PASA) | 90 minutes after oxytocin/placebo application at Visit 3
  Perceived stress will be assessed using the Primary Appraisal secondary Appraisal Scale (PASA) at separate time points before and after Oxytocin Administration using the AUQ at Visit 3 and Visit 4
Primary Appraisal secondary Appraisal Scale (PASA) | 85 minutes after oxytocin/placebo application, i.e. directly fMRI session at Visit 4
  Perceived stress will be assessed using the Primary Appraisal secondary Appraisal Scale (PASA) at separate time points before and after Oxytocin Administration using the AUQ at Visit 3 and Visit 4
Positive and Negative Affect Schedule (PANAS) | 60 minutes after oxytocin/placebo application at Visit 3
  Positive and Negative Affect will be assessed using the Positive and Negative Affect Schedule (PANAS) at separate time points before and after Oxytocin Administration using the AUQ at Visit 3 and Visit 4
Positive and Negative Affect Schedule (PANAS) | 85 minutes after oxytocin/placebo application, i.e. directly fMRI session at Visit 4
  Positive and Negative Affect will be assessed using the Positive and Negative Affect Schedule (PANAS) at separate time points before and after Oxytocin Administration using the AUQ at Visit 3 and Visit 4
Cortisol | 65 minutes after oxytocin/placebo application at Visit 3
  Cortisol plasma levels will be determined using validated Enzyme-linked Immunosorbent Assay (ELISA) methods by the central laboratory at visit 3 after Oxytocin/Placebo administration
Oxytocin | 30 minutes after oxytocin/placebo application at Visit 3
  Oxytocin plasma levels will be determined using validated ELISA methods by the central laboratory at visit 3 after Oxytocin/Placebo administration
Oxytocin | 65 minutes after oxytocin/placebo application at Visit 3
  Oxytocin plasma levels will be determined using validated ELISA methods by the central laboratory at visit 3 after Oxytocin/Placebo administration
Alcohol Cue-induced neural brain activation during an Alcohol cue-reactivity functional magnetic resonance imaging (fMRI) task | During fMRI session at Visit 4, i.e. 40 to 85 minutes after Oxytocin/Placebo administration
  Neural brain activation in the mesocorticolimbic system (whole-brain and Region-of-Interest Analyses (ROIs): ventral striatum, dorsal striatum, insula), measured using the blood oxygenated level dependent (BOLD) response, during presentation of alcohol cues will serve as secondary outcome
Neural Activation during a natural reward cue-reactivity fMRI task | During fMRI session at Visit 4, i.e. 40 to 85 minutes after Oxytocin/Placebo administration
  Neural brain activation in the mesocorticolimbic system (whole-brain and ROIs: ventral striatum, dorsal striatum, insula), measured using the blood oxygenated level dependent (BOLD) response during the presentation of natural reward cues will serve as secondary outcome
Neural Activation during a Face-matching fMRI task | During fMRI session at Visit 4, i.e. 40 to 85 minutes after Oxytocin/Placebo administration
  Neural brain activation in the mesocorticolimbic system (whole-brain and ROIs: ventral striatum, dorsal striatum, insula, amygdala), measured using the blood oxygenated level dependent (BOLD) response during the presentation of emotional faces and neutral shapes will serve as secondary outcome
Neural Activation during a Stop Signal fMRI Task | During fMRI session at Visit 4, i.e. 40 to 85 minutes after Oxytocin/Placebo administration
  Neural brain activation in the mesocorticolimbic system (whole-brain and ROIs: ventral striatum, dorsal striatum, insula, dlPFC), measured using the blood oxygenated level dependent (BOLD) response during a stop signal fMRI task will serve as secondary outcome
Adverse Events (AEs)/Serious Adverse Events (SAEs) and Discontinuation rate | During Study Visits 1 to 6, including the 90 day (±7 day) follow-up period
  Rate of adverse events, serious adverse events and rate of discontinuation of the study due to an adverse event
Subjective quality of life index | At Visit 5, i.e. 30 days (+/- 7 days) after Visit 3
  Quality of life will be assessed using the WHO-QOL-BREF scores
Subjective quality of life index | At Visit 6, i.e. 90 days (+/- 7 days) after Visit 3
  Quality of life will be assessed using the World Health Organization (WHO) Quality of life assessment (WHO-QOL-BREF) scores
Time to relapse during the follow-up period of 90 days (+/- 7 days) | During 90-day (± 7 days) Follow-up
  Time from randomization to relapse to alcohol use (in days)
Cumulative alcohol consumption during the follow-up period of 90 days (+/- 7 days) | During 90-day (± 7 days) Follow-up
  Self-reported cumulative alcohol use (in gram)
Percent heavy drinking days during the follow-up period of 90 days (+/- 7 days) | During 90-day (± 7 days) Follow-up
  Self-reported percent heavy drinking days (in %)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Bach, MD, Study Director — Central Institute of Mental Health, Mannheim
Locations (1):
- Central Institute of Mental Health, Mannheim, Germany

IPD SHARING:
Plan to Share IPD: Yes
Individual de-identified data will be shared, specifically individual participant data that underlie the results of the trial (i.e. primary outcome data [AUQ scores]) will be made available with a respective data dictionary. Secondary Outcome data (e.g. fMRI data) will be made available on aggregated group level (e.g. for the purpose of meta-analyses). Related documents, specifically the study protocol, statistical analysis plan and analytic code will be shared in open-access online repositories. Aggregated data will be made available to publicly accessible repositories (Neurosynth.org), e.g. for the purpose of meta-analyses.
Supporting Information: Study Protocol, SAP
Time Frame: Data will be available upon publication of the results until 3 years after that.
Access Criteria: Individual data will be shared with researchers who provide a methodologically sound proposal (sent to the Principal Investigator/Study Chair of the Trial).

REFERENCES:
- [Derived] Zimmermann S, Thomas BC, Krisam J, Limprecht R, Klose C, Stenger M, Pourbaix M, Ries M, Vollstaedt-Klein S, Koopmann A, Lenz B, Kiefer F, Bach P. ON-ICE trial: Investigation of the combined effects of oxytocin and naltrexone on stress-induced and alcohol cue-induced craving in alcohol use disorder-Study protocol of a phase II randomised double-blind placebo-controlled parallel-group trial. BMJ Open. 2022 Apr 11;12(4):e059672. doi: 10.1136/bmjopen-2021-059672. PMID 35410938